CLINICAL TRIAL: NCT00159692
Title: A Multi-Center, Randomized, Double-Blind, Double-Dummy Study Evaluating The Safety and Efficacy Of The Addition Of Amlodipine To Quinapril Or Losartan In The Treatment Of Diabetic Hypertensive Subjects
Brief Title: Amlodipine Diabetic Hypertension Efficacy Response Trial
Acronym: ADHERE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: A0531063
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Amlodipine

INTERVENTIONS:
Drug: Amlodipine

SUMMARY:
To evaluate the percentage of subjects that reach the diabetic hypertensive blood pressure goal of <130/80 with amlodipine versus placebo in subjects initially treated with quinapril or losartan.

ELIGIBILITY:
Inclusion Criteria:

* Documented evidence of Type 2 diabetes as defined by the ADA guidelines and documented evidence of Hypertension (various SBP/DBP ranges).

Exclusion Criteria:

* A previous history or intolerance or hypersensitivity to calcium channel blockers, ARBs or ACE inhibitors.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 739 (Actual)
Dates: Start 2003-03; Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
The percentage of subjects that reach the JNC diabetic hypertensive BP goal of <130/80 will be assessed at Week 0 (Visit 2-Randomization), Week 5 (Visit 3), Week 9 (Visit 4), Week 15 (Visit 5) and Week 20 (Visit 6 - Final Evaluation).

SECONDARY OUTCOMES:
Percentage of subjects at SBP goal of <130 mmHg and DBP goal of <80mmHg; change from baseline blood pressures (SBP and DBP); percentage of subjects with SBP >160mmHg and/or DBP >100mmHg at Visits 2, 3, 4, 5, 6.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer